CLINICAL TRIAL: NCT06967181
Title: A Phase 1 Trial of CVM150 and CVM26 Intranasal Mumps Virus Vaccines in Healthy Adults
Brief Title: A Phase 1 Trial of Intranasal Mumps Virus Vaccines in Healthy Adults
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: CyanVac LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CVXMV-003
Record Dates: First submitted 2025-05-01; First posted 2025-05-13 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-12

CONDITIONS: Mumps
MeSH Terms: conditions — Mumps

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- CVM150 (Experimental): CVM150: Live PIV5-based MuV vaccine expressing the MuV (Iowa strain/2006) F and HN proteins formulated in 1x sucrose phosphate glutamate ([SPG]; sucrose, KH2PO4, K2HPO4 and L-glutamic acid) buffer.
  Interventions: Biological: CVM150
- CVM26 (Experimental): CVM26: A live, attenuated MuV vaccine based on Iowa strain genetically edited to remove the V and SH protein expression. Formulated in 1x sucrose phosphate glutamate ([SPG]; sucrose, KH2PO4, K2HPO4 and L-glutamic acid) buffer.
  Interventions: Biological: CVM26
- Placebo (Placebo Comparator): Placebo: 0.9% normal sterile saline (purchased commercially).
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: CVM150 — CVM150- Live PIV5-based MuV vaccine expressing the MuV (Iowa strain/2006) F and HN proteins formulated in 1x sucrose phosphate glutamate ([SPG]; sucrose, KH2PO4, K2HPO4 and L-glutamic acid) buffer.
  Arms: CVM150
Biological: CVM26 — CVM26: A live, attenuated MuV vaccine based on Iowa strain genetically edited to remove the V and SH protein expression. Formulated in 1x sucrose phosphate glutamate ([SPG]; sucrose, KH2PO4, K2HPO4 and L-glutamic acid) buffer.
  Arms: CVM26
Other: Placebo — Placebo: 0.9% normal sterile saline (purchased commercially).
  Arms: Placebo

SUMMARY:
The purpose of this trial is to evaluate the safety and immunogenicity of CVM150 and CVM26. The trial will enroll up to 60 healthy participants.

DETAILED DESCRIPTION:
This is a randomized, blinded, placebo-controlled, phase 1 clinical trial to evaluate the safety and immunogenicity of CVM150 and CVM26 in healthy adults who received the recommended 2 doses of mumps vaccine (as measles-mumps-rubella [MMR] or MMR -varicella [MMRV]) in childhood.

Number of Participants:

A total of up to 60 participants, aged 18-29 years, are planned to be enrolled.

Treatment Assignment: All participants will be randomized to receive a single intranasal dose of CVM150, CVM26 or intranasal saline placebo (1:1:1) on Day 1.

Study visits: Participants will be asked to complete approximately 6-8 clinic visits, over a period of approximately 12 months duration per participant.

ELIGIBILITY:
Inclusion Criteria:

* Individuals ≥18 years and <30 years of age at the time of consent.
* Willing and able to comply with all scheduled visits, vaccination plan, laboratory tests and other trial procedures.
* Determined by medical history, complete physical examination and clinical judgement of the investigator to be in good state of health*.

  * As determined by medical history and physical examination to evaluate acute or ongoing chronic medical diagnoses/conditions that have been present for at least 90 days, which would affect the safety assessment of subjects. Chronic medical diagnoses/conditions should be stable for the last 60 days (no hospitalizations, emergency room (ER), or urgent care for condition or need for supplemental oxygen). This includes no change in chronic prescription medication, dose, or frequency due to deterioration of the chronic medical diagnosis/condition in the 60 days before enrollment. Any prescription change that is due to change of health care provider, insurance company, etc., or done for financial reasons, and in the same class of medication, will not be considered a deviation of this inclusion criterion.

Any change in prescription medication due to improvement of a disease outcome, as determined by the participating site principal investigator (PI) or appropriate sub- investigator, will not be considered a deviation of this inclusion criterion. Subjects may be on chronic or as needed (prn) medications if, in the opinion of the participating site PI or appropriate sub-investigator, they pose no additional risk to subject safety or assessment of reactogenicity and immunogenicity, and do not indicate a worsening of medical diagnosis/condition. Similarly, medication changes subsequent to enrollment and trial vaccination are acceptable provided the change was not precipitated by deterioration in the chronic medical condition, and there is no anticipated additional risk to the subject or interference with the evaluation of responses to trial vaccination.

* Prior receipt of two doses of mumps vaccine in childhood (as MMR or MMRV).
* Women of childbearing potential* must agree to use or have practiced true abstinence** or use at least one acceptable primary form of contraception.***, **** Note: These criteria are applicable to females in a heterosexual relationship and child-bearing potential (i.e., the criteria do not apply to subjects in a same sex relationship).

  *Not of childbearing potential: post-menopausal females (defined as having a history of amenorrhea for at least one year) or a documented status as being surgically sterile (hysterectomy, bilateral oophorectomy, tubal ligation/salpingectomy, or Essure® placement).

  **True abstinence is no sexual intercourse 100% of the time (i.e. male's penis never enters the female's vagina). Periodic abstinence (e.g., calendar, ovulation, symptothermal, post- ovulation methods) and withdrawal are not acceptable methods of contraception.

  ***Acceptable forms of primary contraception include monogamous relationship with a vasectomized partner who has been vasectomized for 180 days or more prior to the subject's vaccination, intrauterine devices, birth control pills, and injectable/implantable/insertable hormonal birth control products, condom, or diaphragm with spermicide. If barrier methods are to be used, then double barrier methods of protection are required, i.e. male condom, in combination with a cap, diaphragm, or sponge with spermicide.

  ****Must use at least one acceptable primary form of contraception for at least 28 days prior to vaccination and at least one acceptable primary form of contraception for 90 days after last vaccination. If barrier methods are to be used, then double barrier methods of protection are required, i.e. male condom, in combination with a cap, diaphragm, or sponge with spermicide.
* Women of childbearing potential must have a negative urine or serum pregnancy test within 24 hours prior to vaccination.
* Male subjects of childbearing potential* must use condoms to ensure effective contraception with a female partner of childbearing potential from vaccination until 90 days after vaccination. Such female partners must also use an acceptable form of primary contraception as described under inclusion criterion #5. If barrier methods are to be used, then double barrier methods of protection are required, i.e. male condom, in combination with a cap, diaphragm, or sponge with spermicide.

  *Biological males who are post-pubertal and considered fertile until permanently sterile by bilateral orchiectomy or vasectomy.
* Female subjects agree to refrain from egg donation from time of vaccination until 90 days after vaccination.
* Male subjects agree to refrain from sperm donation from the time of vaccination until 90 days after vaccination.

Exclusion Criteria:

* Mumps vaccination within 10 years.
* History of mumps virus infection.
* History of parotitis, epididymoorchitis or oophoritis.
* COVID-19 infection <30 days prior to planned trial vaccine administration.
* Influenza infection < 30 days prior to planned trial vaccine administration.
* Pregnant or breastfeeding participants.
* History of severe respiratory infection (e.g., need for oxygenation or ventilatory support).
* Any prior receipt of a PIV5-based vaccine (e.g., CVXGA [an intranasal COVID-19 vaccine] or BLB-201 [an intranasal RSV vaccine] being developed by CyanVac/Blue Lake Biotechnology).
* Any prior receipt of an investigational mumps vaccine.
* Chronic rhinitis, nasal septal defect causing significant breathing problems, cleft palate, nasal polyps, or other nasal abnormality that might affect vaccine administration.
* Current or planned simultaneous participation in another interventional trial or receipt of any investigational trial product within 28 days prior to trial vaccine administration.
* A history of anaphylaxis, urticaria, or other significant adverse reaction requiring medical intervention after receipt of a vaccine (licensed or unlicensed).
* A history of meningitis, encephalitis, facial palsy, Guillain-Barré syndrome, or transverse myelitis.
* Cochlear implants or history of cerebrospinal fluid leak or active communication between the cerebrospinal fluid (CSF) and oropharynx, nasopharynx, nose or ear.
* A history of myocarditis or pericarditis at any time prior to enrollment, history of Kawasaki disease, or history of multisystem inflammatory syndrome after COVID-19 infection.
* Received or plans to receive an inactivated vaccine within 14 days prior to or after trial vaccine.
* Received or plans to receive a live virus vaccine within 28 days prior to or after trial vaccine.
* Bleeding disorder diagnosed by a healthcare provider (e.g., factor deficiency, coagulopathy, or platelet disorder requiring special precautions) or bleeding difficulties with intramuscular injections or blood draws.
* Current or previous diagnosis of a significant immunocompromising condition or other immunosuppressive condition.
* Resides with someone who is severely immunocompromised.
* Advanced liver or kidney diseases.
* HIV infection, active Hepatitis B virus infection, history of positive serology for Hepatitis C.
* Received oral, intramuscular, or intravenous systemic immunosuppressants, or immune-modifying drugs for >14 days in total within 6 months prior to administration of trial vaccine (for corticosteroids > / = 20 mg/day of prednisone equivalent).
* History of significant/severe wheeze, respiratory symptoms resulting in hospitalization, or known bronchial hyperreactivity to viruses.
* Received immunoglobulin or blood-derived products, within 3 months prior to trial vaccine dose.
* Received chemotherapy, immunotherapy, or radiation therapy within 6 months prior to trial vaccine dose.
* Trial personnel or an immediate family member or household member of trial personnel.
* Is acutely ill or febrile 72 hours prior to or at vaccine dosing day (fever defined as > / = 38.0°C/100.4°F). Subjects meeting this criterion may be rescheduled within the relevant window periods but may require screening for respiratory pathogen infection.
* Receipt or anticipated receipt of, within 7 days prior to through 28 days after trial vaccination, any intranasal medication including FDA-approved prescription or over-the-counter products or non-FDA-approved alternative medicine products (e.g., Ayurvedic oil or other naturopathic substances).
* Currently smoking or vaping, or history of regular smoking or vaping in the past two years (average of 1 cigarette or equivalent daily).
* Active alcohol use disorder or alcohol abuse or active illicit drug abuse.
* Anticipated use of nasal irrigation (e.g., Neti Pot™) after enrollment through 28 days after trial vaccination.
* Nasal piercing within 30 days prior to trial vaccination or planned 30 days after trial vaccination.

Ages: 18 Years to 29 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2025-05-14 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
The percentage of participants who experience any solicited local reactogenicity symptom pertaining to intranasal administration through 7 days post-vaccination (Day 1 through Day 8) | Day 1 through Day 8
  The percentage of participants who experience any solicited local reactogenicity symptom pertaining to intranasal administration through 7 days post-vaccination (Day 1 through Day 8)
The percentage of participants who experience any solicited systemic reactogenicity symptom through 7 days postvaccination (Day 1 through Day 8) | Day 1 through Day 8
  The percentage of participants who experience any solicited systemic reactogenicity symptom through 7 days postvaccination (Day 1 through Day 8)
The percentage of participants who experience any unsolicited adverse event (AE) through 28 days post-vaccination (Day 1 through Day 29) | Day 1 through Day 29
  The percentage of participants who experience any unsolicited adverse event (AE) through 28 days post-vaccination (Day 1 through Day 29)
The percentage of participants who experience the following events through 6 months post-vaccination: • SAEs • MAAEs • AESIs • NOCMCs | Day 1 through Day 181
  The percentage of participants who experience the following events through 6 months post-vaccination:
  * serious adverse events (SAEs)
  * medically attended adverse events (MAAEs)
  * adverse events of special interest (AESIs)
  * new onset chronic medical conditions (NOCMCs)
The percentage of participants who experience the following events through 12 months post-vaccination: • SAEs • MAAEs • AESIs • NOCMCs | Day 1 through Day 366
  The percentage of participants who experience the following events through 12 months post-vaccination:
  * serious adverse events (SAEs)
  * medically attended adverse events (MAAEs)
  * adverse events of special interest (AESIs)
  * new onset chronic medical conditions (NOCMCs)

SECONDARY OUTCOMES:
Geometric mean fold rise (GMFR) of serum mumps virus (MuV) neutralizing antibodies (nAbs) on Day 15 and/or Day 29 | Day 15 and/or Day 29
  Geometric mean fold rise (GMFR) of serum mumps virus (MuV) neutralizing antibodies (nAbs) on Day 15 and/or Day 29
Proportion of participants with an increase in serum MuV-specific immunoglobulin G (IgG) antibodies (by enzyme-linked immunosorbent assay [ELISA]) at Day 15 and/or Day 29 | Day 15 and/or Day 29
  Proportion of participants with an increase in serum MuV-specific immunoglobulin G (IgG) antibodies (by enzyme-linked immunosorbent assay [ELISA]) at Day 15 and/or Day 29
Proportion of participants with an increase in MuV-specific cell mediated immune responses (CMI) in PBMCs at Day 8, 15 and/or Day 29 | Day 8, Day 15 and/or Day 29
  Proportion of participants with an increase in MuV-specific cell mediated immune responses (CMI) in PBMCs at Day 8, 15 and/or Day 29
Proportion of participants with an increase in mucosal (nasal and/or saliva) MuV- specific IgA at Day 15 and/or Day 29 | Day 15 and/or Day 29
  Proportion of participants with an increase in mucosal (nasal and/or saliva) MuV- specific IgA at Day 15 and/or Day 29
Assess duration of vaccine virus shedding after vaccination | Day 1 through Day 29
  Assess duration of vaccine virus shedding after vaccination

CONTACTS AND LOCATIONS:
Overall Officials: Hong Jin, Study Chair — CyanVac LLC
Locations (3):
- United States (3):
  - University Of Rochester Medical Center, Rochester, New York
  - Cincinnati Children's Hospital Medical Center Vaccine Research Center, Cincinnati, Ohio
  - Coastal Carolina Research Center, North Charleston, South Carolina

IPD SHARING:
Plan to Share IPD: No